CLINICAL TRIAL: NCT01124825
Title: Use of New Supraglottic Airway Devices in Severely Obese Patients: A Feasibility Study
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: No subjects enrolled. Funding withdrawn by sponsor.
Sponsor: University of Louisville (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: UofL IRB #09.0619
Record Dates: First submitted 2010-05-12; First posted 2010-05-17 (Estimated); Last update posted 2012-11-14 (Estimated); Status verified 2012-11

CONDITIONS: Obesity
Keywords: Anesthesia induction and maintenance; Surgery
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- IGel (Active Comparator): Subjects will receive an IGel(TM) airway induction and maintenance of positive pressure ventilation
  Interventions: Device: IGEL
- King Airway (Active Comparator): Subject will receive a KING-LTS-D(TM) for induction and maintenance of positive pressure ventilation
  Interventions: Device: King airway

INTERVENTIONS:
Device: IGEL — iGEL(TM) airway will be used for induction and maintenance of positive pressure ventilation
  Arms: IGel
Device: King airway — KING-LTS-D(TM) airway will be used for induction and maintenance of positive pressure ventilation
  Arms: King Airway

SUMMARY:
The purpose of this study is to determine whether two new airway devices used during anesthesia called iGEL™ and KING-LTS-DTM work well and are safe in obese patients. They both work well in thin patients, but have not been tested in obese patients.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for elective surgery with an estimated duration of 30 to 120 minutes
* American Society of Anesthesiologists (ASA) status I-III
* Aged 18 to 65 years.
* Body mass index (BMI) ≥ 35 kg/m2

Exclusion Criteria:

* A history of difficult intubation;
* Immobilized cervical spine;
* Oxygen saturation less than 95% at room air;
* A history of uncontrolled gastroesophageal reflux or hiatus hernia;
* A history of ulcer surgery including vagotomy;
* Previous gastric bypass surgery;
* Diabetic gastroparesis;
* Patients with known coagulation disorders (e.g. hemophilias, von Willebrand disease, factor V leiden diseases) or on systemic anticoagulation drugs (e.g. continuous heparin infusion); Patients with abnormal coagulation tests will be also excluded. However, asymptomatic patients will not be tested on any coagulation disorders.
* Any pathologies of the mouth, pharynx or larynx, the access to the airway is restricted, or a difficult tracheal intubation is anticipated.
* Pregnant or breast-feeding (pregnancy status will be confirmed by a pregnancy test, as it is standard for all surgical procedures at the University hospital).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-07; Primary Completion 2012-05 (Estimated); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Airway Sealing Pressure | 1-3 hours
  Oropharyngeal leak pressure in cm H2O for the duration of the case at 1, 15, 30, 60, 120 minutes.

SECONDARY OUTCOMES:
Difference in insertion time for one of the supraglottic airway devices | 1-3 hours
  Effective airway time (time required to place the endotracheal tube/ supraglottic airway device).

CONTACTS AND LOCATIONS:
Overall Officials: Detlef Obal, MD, Principal Investigator — University of Louisville
Locations (1):
- University of Louisville Hospital, Louisville, Kentucky, United States

REFERENCES:
- [Background] Kheterpal S, Martin L, Shanks AM, Tremper KK. Prediction and outcomes of impossible mask ventilation: a review of 50,000 anesthetics. Anesthesiology. 2009 Apr;110(4):891-7. doi: 10.1097/ALN.0b013e31819b5b87. PMID 19293691